CLINICAL TRIAL: NCT06211959
Title: Evaluating the Effectiveness of Implementation Intentions to Strengthen Approach-avoidance Training : Pilot Study on Alcohol Use Disorder
Brief Title: Evaluating the Effectiveness of Implementation Intentions to Strengthen Approach-avoidance Training
Acronym: IMBA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique de la Mitterie (Other)
Responsible Party: Principal Investigator, Michaël RACODON, Head of clinical research, Clinique de la Mitterie
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A02415-34
Record Dates: First submitted 2023-12-26; First posted 2024-01-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
Keywords: cognitive bias; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: single-centre, randomised, superiority study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Classical Approach Bias Modification (Experimental): The 3 arms will follow a similar procedure, except that they will receive 3 different experimental interventions, dependly on their conditions.
  Interventions: Behavioral: Approach Bias Modification with Implementation Intentions
- Approach Bias Modification with Implementation Intentions (Experimental): The 3 arms will follow a similar procedure, except that they will receive 3 different experimental interventions, dependly on their conditions.
  Interventions: Behavioral: Approach Bias Modification with Implementation Intentions
- Sham-training (Placebo Comparator): The 3 arms will follow a similar procedure, except that they will receive 3 different experimental interventions, dependly on their conditions.
  Interventions: Behavioral: Approach Bias Modification with Implementation Intentions

INTERVENTIONS:
Behavioral: Approach Bias Modification with Implementation Intentions — Participants in each experimental condition will perform different variants of the Approach-Avoidance Task (i.e., a task that is widely used in the litterature to assess and modify the approach bias toward alcohol - the relative ease to approach alcohol rather than to avoid it). Participants in the classical Approach Bias Modification conditions will perform a version of this task which will train them to (almost-)systematically emit an avoidance response toward alcohol ; Participants in the Approach Bias Modification with Implementation Intentions condition will perform the same version of the task but will additionnaly have to complete a planning intervention (i.e., implementation intentions) to help them avoiding alcohol; Participants in the Sham-training condition will perform a version of this task which require them to approach alcohol as often as they have to avoid it (i.e., no real training).
  Other Names: Classical Approach Bias Modification

SUMMARY:
Approach Bias Modifcation corresponds to computerized interventions designed to change a cognitive bias (i.e., the approach bias) that may contribute to the maintenance of Alcohol Use Disorder. This study aims to compare the effectiveness of a classical Approach Bias Modification program, an Approach Bias Modification program integrating a planning strategy (i.e., implementation intentions) and a Sham-training to decrease the approach bias (from pre to post-test), and Alcohol Use Disorder symptomatology (from baseline to follow-up). 112 patients will be recruited for this study.

DETAILED DESCRIPTION:
The Approach Bias is considered to be a maintenance factor of Alcohol Use Disorder. It correspond to the relative ease to approach alcohol rather than to avoid it. Approach Bias Modifcation correspond to computerized interventiond designed to change it by training participants to emit avoidance response (e.g., pull the joystick away) toward alcohol stimuli (e.g., alcohol pictures). Those programs have shown their effectiveness to promote abstinence among Alcohol Use Disorder patients. This study aims to compare the effectiveness of a classical Approach Bias Modification program to the one of a similar program integrating a planning add-on strategy named implementation intentions and to a Sham-training. 112 patients will be recruited for this study at Clinic de la Mitterie rehab center. During their hospitalization, participants will have to complete: a baseline that assess Alcohol Use Disorder symptomatology (i.e., alcohol consumption, alcohol consumption, and alcohol-related consequences) and other alcohol-related variables (e.g., motivation and self-efficacy), a pre-test that assess the approach bias, 6 sessions of one of the three experimental interventions {classical Approach Bias Modification, Approach Bias Modification with Implementation Intentions, Sham-training}, and a post-test that reassess the approach bias. After their hospitalization, they will have to complete a 2, 4 and 6-month online follow-up that reasses Alcohol Use Disorder symptomatology. It is expect that the Approach Bias Modification program with implementation intentions will decrease the approach bias and Alcohol Use Disorder symptomatology more than the classical program, that will also decrease it more than the Sham-training.

ELIGIBILITY:
Inclusion Criteria:

* care at the clinic for Alcohol Use Disorder,
* have an e-mail address,
* written and spoken French,
* signing informed consent.

Exclusion Criteria:

* not currently remissioned for the Alcohol Use Disorder,
* no other Substance Use Disorder (except tobaco one)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
Approach-Avoidance Task (AAT) | 2 weeks
  The approach bias toward alcohol

SECONDARY OUTCOMES:
Alcohol consumption | 2 weeks
  The Alcohol Use Disorder Identification Test - Consumption (AUDIT)

OTHER OUTCOMES:
Alcohol dependence | 2 weeks
  The Short Alcohol Dependence Data questionnaire (SAAD)
Alcohol-related consequences | 2 weeks
  The Short Inventory of Problems - Revised (SIP-R)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique la Mitterie, Lille, France

IPD SHARING:
Plan to Share IPD: Yes
1. sign an informed consent and to complete a baseline that assess the secondary outcomes measures as well as other alcohol-related measures (e.g., motivation and self-efficacy to change alcohol consumption).
  2. complete a pre-test that asssess the primary outcome measure (i.e., the approach bias).
  3. receive 6 session of their respective experimental intervention
  4. complete a post-test to reassess the primary outcome measure (i.e., the approach bias).
  Follow-up Phase. After participants hospitalization, participants will have to complete a 2, 4, and 6-month online follow-up that reassess the secondary outcome measures (i.e., alcohol consumption, alcohol dependence, and alcohol-related-consequences).
Supporting Information: Study Protocol